## IVROP ReadyforLIFE Program Evaluation Statistical Analysis Plan

August 29, 2024

ClinicalTrials.gov ID: NCT05244447

## Analysis approach

The main goal of this descriptive study is to assess pre-post change scores in the means of the outcome constructs listed above among program participants before, immediately following, and one year after primary workshops. We will use paired sample t-tests to assess the magnitude and significance of mean score changes among program participants in the analytic sample for each outcome.

The analytic sample for each outcome construct consists of study participants who have a non-missing value at baseline and follow-up time points for that outcome (complete case). The analytic sample may vary by outcome construct based on prevalence of missing data at the baseline, post, or follow-up surveys for those questions. The final report will include descriptive statistics about the sample for each outcome, including which optional services (2.0, PLUS, or none) that participants received. As mentioned in the Outcomes section above, a respondent who answers some but not all survey items in a given outcome construct matrix will have their outcome value assigned as missing if they do not respond to at least 80% of the items in the construct. We will not impute missing baseline or outcome data for our analyses. Findings are considered statistically significant based on p < 0.05, two-tailed test. We will adjust our p-values for multiple hypothesis testing and report the adjusted p-values in the appendix of the final report.

As part of data preparation and cleaning, we will check for inconsistent and seemingly inaccurate data. The largest source of potentially inconsistent data that we anticipate is duplicate local evaluation surveys. Participants are able to, and occasionally do, retake the local evaluation surveys on Qualtrics. In the case of duplicate survey data, where participants have taken a local evaluation survey more than one time, we plan to take the following approach:

- Check for incorrectly entered Client IDs that inaccurately flag surveys as duplicates. Using the name and/or DOB fields on the local evaluation survey, we will check that responses that appear to be duplicates were in fact collected from the same participant multiple times (i.e., are true duplicates).
   If not, we will correct Client IDs as necessary.
- Check for completeness. If one duplicate survey is complete while the other is not, we will use the most complete survey to minimize item non-response.
- If both duplicate surveys are equally complete, we will use the first response that a participant submitted, as indicated by the Recorded Date field on the Qualtrics data export.

Raw data sets for baseline, exit, and follow-up survey data will be cleaned and prepared for analyses using the R Studio statistical software package. nFORM survey responses and will be downloaded using the Data Export feature of nFORM, and local evaluation survey responses will be exported from Qualtrics. All exports will be imported into R and cleaned separately before data sets are merged into a final, wide format file for analyses using nFORM Client ID as the unique identifier for matching observations.

As a sensitivity check, we plan to repeat the analyses using only participants who received primary workshops (i.e., excluding 2.0 and PLUS participants).

## Attrition

The ReadyforLIFE program has consistently exceeded its post-survey and follow-up data collection

participation targets, which has helped to reduce overall sample attrition. This success has been due in large part to strong program completion rates and the follow-up collection strategies that both program and evaluation staff have used with youth participants. Facilitators and life coaches explain the importance of the evaluation at the beginning of the program and inform youth that they will be eligible for a \$50 incentive (a Giftogram gift card redeemable at either Walmart or Target) if they complete the 1-year follow-up survey. This message was reinforced by program alumni in schools who verified that they received their incentives after completing the survey.

Midwest Evaluation and Research employs a dedicated survey tracking team that begins reaching out to eligible participants one month before their 1-year follow-up survey is due, using the contact information collected by program staff during the enrollment process. Participants are eligible for a follow-up survey if they have parental consent and youth assent to be part of the study and have completed at least one baseline survey, regardless of program completion status or program delivery format. The survey tracking team uses multiple methods of contact (text, email, phone calls, letters, and social media) to reach participants. Youth can take the 1-year follow-up survey online (using a link provided via text, email, or social media, or using a QR code provided via letter), or they can opt to complete a survey over the phone with a survey tracking team member.

Sample attrition is tracked on an ongoing basis as part of the bi-weekly Continuous Quality Improvement (CQI) team meetings that MER and IVROP attend together. If response rates drop below the target of 70%, interventions would be put in place to try to increase response rates; however, this has not been necessary to date, as follow-up response rates are currently over 80%.

At the outcome level, attrition will be reported descriptively in the final report. For each outcome construct, we plan to report the proportion of the sample that is missing for that outcome measure and for what reason (e.g., survey non-response, skipped items, exceeded 20% threshold for item missingness within a construct). We will report descriptive statistics for baseline responses, gender as reported on the Applicant Characteristics Survey (ACS), and age as reported on the ACS to compare those who are and are not in the sample for each outcome.